CLINICAL TRIAL: NCT02926469
Title: Virtual Reality Analgesia in Labor: The VRAIL Pilot Study
Acronym: VRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Melissa Bauer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00116129
Record Dates: First submitted 2016-09-14; First posted 2016-10-06 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Labor Pain
Keywords: Virtual Reality; Analgesia; Immersive Virtual Reality; VR; Labor; Pain
MeSH Terms: conditions — Labor Pain; Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): For patients presenting in labor and desiring standard care (natural childbirth without pain medications, systematic distraction, or alternative therapies) the patient will experience their contractions. Afterwards they will answer pain and anxiety questionnaires.
- Virtual Reality (Experimental): For patients presenting in labor and desiring standard care (natural childbirth without pain medications, systematic distraction, or alternative therapies) the patient will experience their contractions while using immersive Virtual Reality.Afterwards they will answer pain and anxiety questionnaires.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Using Virtual Reality during labor
  Arms: Virtual Reality

SUMMARY:
The purpose of the proposed study is to evaluate the feasibility of using immersive Virtual Reality (VR) during labor. We will also explore whether VR distraction is helpful for reducing subjective pain during labor, even if this pain is severe or excruciating. We predict that VR is feasible in this setting and that VR distraction will reduce acute pain and anxiety during labor.

DETAILED DESCRIPTION:
This study used an over the counter consumer product to create a virtual reality experience so that we could assess whether there was a decrease in perception of pain.

ELIGIBILITY:
Inclusion Criteria:

* Any woman giving birth for the first time at or after 32 weeks
* Low risk pregnancy without obstetric complications
* In first stage of labor for vaginal delivery
* Desires non-pharmacologic alternative for pain control

Exclusion Criteria:

* Younger than 18 or older than 45 years of age
* Presence of fetal or placental anomaly
* High risk pregnancy or anesthetic concerns (BMI>40, difficult airway, hemorrhage, nonreassuring FHR, malpresentation)
* Current use of pharmacologic analgesia including neuraxial anesthesia
* Not capable of answering study measures using numeric rating scale
* Any face/head/neck injuries that interfere with the use of Virtual Reality equipment
* Any form of contact precautions
* Severe hearing or vision deficits
* Susceptibility to motion sickness
* Seizure history
* History of psychiatric disorder, chronic pain, migraines, or addiction
* Delirium, psychosis, any form of developmental delay, or Organic Brain Disorder
* Requiring an interpreter for communication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Pain and Anxiety | one time for the duration of one minute after 10 minutes of contractions with standard care
  Pain is measured one time after 10 minutes of contractions with standard care, by asking the subjects about their pain and anxiety level, using a questionnaire called graphic rating scale.
Pain and Anxiety | one time for the duration of one minute after 10 minutes of contractions using Virtual Reality
  Pain is measured one time after 10 minutes of contractions with Virtual Reality, by asking the subjects about their pain and anxiety level, using a questionnaire called graphic rating scale.
Satisfaction | one time for the duration of one minute after using Virtual Reality
  Evaluate women's attitudes towards Virtual Reality use during labor through a satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bauer, DO, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Von Voigtlander Women's Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frey DP, Bauer ME, Bell CL, Low LK, Hassett AL, Cassidy RB, Boyer KD, Sharar SR. Virtual Reality Analgesia in Labor: The VRAIL Pilot Study-A Preliminary Randomized Controlled Trial Suggesting Benefit of Immersive Virtual Reality Analgesia in Unmedicated Laboring Women. Anesth Analg. 2019 Jun;128(6):e93-e96. doi: 10.1213/ANE.0000000000003649. PMID 31094789